CLINICAL TRIAL: NCT06036901
Title: Assessment of Coronary Artery Disease in Asymptomatic Population Undergoing Coronary Computed Tomography Angiography: A Single Center, Prospective Observational Study
Brief Title: Asan Medical Center CCTA Registry
Status: Completed | Type: Observational
Sponsor: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Principal Investigator, Seung-Whan Lee, Principal investigator, clinical professor, CardioVascular Research Foundation, Korea
Other Study IDs: CardioVascularRF
Record Dates: First submitted 2023-08-15; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Risk Factor; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary CT — Coronary CT evaluation

SUMMARY:
A total of 9269 adults who received CCTA scans for coronary disease evaluation during a general medical checkup at the Health Screening and Promotion Center in Asan Medical Center, Seoul, Korea between January 2007 and December 2011 were initially selected. All participants were provided with information about the potential benefits and risks of CCTA and made the decision to undergo the procedure at their own expense. They were also informed that their clinical and radiological data would be used for this study and gave their consent. Of these individuals, 7129 agreed to participate, and 6343 were enrolled in this CCTA registry.

ELIGIBILITY:
Exclusion Criteria:

1. a previous history of angina or myocardial infarction;
2. abnormal rest electrocardiographic results, i.e., pathological Qwaves, ischemic ST segments or T wave changes, or left bundle-branch blocks;
3. insufficient medical records;
4. structural heart diseases;
5. a prior history of open heart surgery or percutaneous coronary intervention;
6. a previous cardiac procedure; or
7. renal insufficiency (creatinine N1.5 mg/dL)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 20 years and older had undergone self-referral CCTA evaluation as part of a general health examination in the Health Screening and Promotion Center at Asan Medical Center from January 2007 to December 2011.
Sampling Method: Non-Probability Sample
Enrollment: 6343 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The prevalence of CAD | 5 years
  Diameter stenosis >50% in any coronary artery by coronary CT angiography

SECONDARY OUTCOMES:
All cause mortality | 5 years
cardiovascular mortality | 5 years
  any death caused by a cardiovascular problem or if there was no identified cause of death
myocardial infarction | 5 years
  Number of participants with an increase in cardiac enzyme above the upper reference limit with ischemic symptoms or signs.
Revascularization | 5 years
  Number of participants with any percutaneous or surgical revascularization procedure during follow-up.

IPD SHARING:
Plan to Share IPD: No